CLINICAL TRIAL: NCT07364565
Title: The Antiplaque and Antigingivitis Effect of Pure Green Tea Mouth Wash Compared to Placebo and Essential Oils Mouth Washes: A Double Blinded Randomized Controlled Clinical Trial.
Brief Title: The Antiplaque and Antigingivitis Effect of Pure Green Tea Mouth Wash Compared to Placebo and Essential Oils Mouth Washes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Lana Bader, Dr, Assistant Professor, Jordan University of Science and Technology
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 425/2025; 2025/185-1 (Other: Institutional Review Board at Jordan University of Science and Technology)
Record Dates: First submitted 2025-12-29; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Dental Plaque; Patient Reported Outcome; Gingival Inflammation and Bleeding; Gingival Inflammation; Gingival Bleeding; Gingivitis
Keywords: Green tea; Gingival inflammation; Plaque index; Essential oils; Mouthwash; Bleeding on probing; Camellia sinensis; Herbal medicine; Periodontal health
MeSH Terms: conditions — Dental Plaque; Gingivitis; Hemorrhage; Gingival Hemorrhage

STUDY DESIGN:
Intervention Model Description: This is a double-blinded, parallel group, randomised, controlled, clinical trial with four arms: pure green tea mouthwash, Listerine Total Care, Listerine Green Tea, and placebo. Participants will rinse twice daily for three weeks. They will be prohibited from all forms of mechanical plaque control during the study period.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants, investigators, and outcome assessors will be blinded. Mouthwashs will be emptied in opaque bottles. They will be coded and unlabeled. A trained dental assisstant will be responsable about disposing the assigned mouth wash to the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pure Green Tea Mouthwash (Experimental): Participants in this group will use a mouthwash prepared from pure green tea extract. The solution will be brewed by infusing 1 g of green tea leaves in 100 ml of boiling deionized water for 20 minutes, cooled, filtered, and stored in brown glass bottles.
  Interventions: Drug: Pure Green Tea Mouthwash
- Listerine Total Care Mouthwash (Active Comparator): Participants in this group will use Listerine Total Care essential oils mouthwash, containing eucalyptol, menthol, methyl salicylate, and thymol.
  Interventions: Drug: Listerine Total Care Mouthwash
- Listerine Green Tea Mouthwash (Active Comparator): Participants will use Listerine Green Tea mouthwash, an essential oil-based product enhanced with green tea extract.
  Interventions: Drug: Listerine Green Tea Mouthwash
- Placebo Mouthwash (Placebo Comparator): The solution contains only water and additive flavor with no active anti-inflammatory ingredients.
  Interventions: Other: Placebo Mouthwash

INTERVENTIONS:
Drug: Pure Green Tea Mouthwash — Participants in this group will use a mouthwash prepared from pure green tea extract. The solution will be brewed by infusing 1 g of green tea leaves in 100 ml of boiling deionized water for 20 minutes, cooled, filtered, and stored in brown glass bottles. Participants will rinse with 10 ml of the mouthwash twice daily for 30 seconds over 3 weeks. They should not use any form of oral hygiene during the study period.
  Arms: Pure Green Tea Mouthwash
Drug: Listerine Total Care Mouthwash — Participants in this group will use Listerine Total Care essential oils mouthwash, containing eucalyptol, menthol, methyl salicylate, and thymol. All participants will rinse with 10 ml twice daily for 30 seconds for 3 weeks. They should not use any form of oral hygiene during the study period. This will serve as an active control to compare the efficacy of essential oils with the pure green tea formulation and placebo.
  Arms: Listerine Total Care Mouthwash
Drug: Listerine Green Tea Mouthwash — Participants will use Listerine Green Tea mouthwash, an essential oil-based product enhanced with green tea extract and fluoride. All participants will rinse with 10 ml twice daily for 30 seconds over 3 weeks. They should not use any form of oral hygiene during the study period. This will allow comparison between a commercial green tea-containing mouthwash and the pure green tea solution.
  Arms: Listerine Green Tea Mouthwash
Other: Placebo Mouthwash — Participants will rinse with 10 ml of a placebo solution consisting of pure water with a flavored additive to mimic taste and color. They should not use any form of oral hygiene during the study period. The solution contains no active anti-inflammatory ingredients. The placebo serves to determine baseline changes in plaque and gingivitis without active intervention.
  Arms: Placebo Mouthwash

SUMMARY:
The goal of this clinical trial is to to evaluate the antiplaque and antigingivitis effect of pure green tea mouthwash compared to placebo and essential oils mouthwashes in healthy patients.

The main questions it aims to answer are:

* Does pure green tea mouthwash effectively reduce dental plaque?
* Does pure green tea mouthwash reduce gingival inflammation?

Researchers will compare pure green tea mouthwash to Listerine Total Care, Listerine Green Tea, and placebo to see if there is a difference in plaque accumulation and gum inflammation reduction.

Participants will be prohibited from using any sort of oral hygiene parctice for the whole study period (3 weeks). Instead, they will rinse with 10 ml of their assigned mouthwash twice daily for 30 seconds. Plaque index, gingival index, and staining index will be examined at multiple intervals and participants will rate their sense of oral freshness and good breath.

DETAILED DESCRIPTION:
• Study Design

This study will be a double-blinded, randomized, controlled, clinical trial with a parallel group design. Participants will be randomly allocated into four groups:

Group P: placebo (pure water with a flavored additive) solution. Group T1: pure green tea mouthwash. Group T2: Listerine Total Care mouthwash. Group T3: Listerine Green Tea mouthwash.

All participants will be instructed to rinse with 10 ml of the assigned mouthwash for 30 seconds twice daily over a three-week experimental period. The study will follow the experimental gingivitis model, during which participants will refrain from all forms of mechanical plaque control.

* Sample Size A total of 44 dental participants, aged between 18-50 years, will be recruited. Each group will consist of 11 participants, providing a power of 80% to detect a difference of 0.2 in mean plaque index values between groups, with a p-value < 0.05 and a β-error of 20%.
* Ethical Considerations All participants will be informed about the study objectives, methodology, and possible risks. Written informed consent will be obtained before participation. All procedures will follow ethical standards and the principles of the Declaration of Helsinki.
* Data Collection and Clinical Assessments Clinical examinations will be performed at baseline (T0), day 7 (T1), day 14 (T2), and day 21 (T3). The following parameters will be recorded: plaque index, gingival index, staining index, and patients reported outcome in regards to their perciption of freshness and good breath.

After the experimental period (T3), participants will receive a professional cleaning and fluoride application, and will be followed for two additional weeks to ensure the restoration of oral health.

* Randomization and Blinding Randomization will be performed using a computer-generated sequence by an independent researcher. The mouthwash samples will be provided in coded and unlabeled containers to ensure blinding of both participants and the examiner. A third party will be responsible about desposing the assigned mouth wash to the patients.
* Adverse Events Monitoring Participants will be closely monitored throughout the study for any possible adverse effects such as gingival irritation, sensitivity, or allergic reactions. Any incident will be documented and managed according to the study protocol. Any participant who experience an adverse event will be excluded from the study.

ELIGIBILITY:
Inclusion criteria:

* Non-smokers
* Systemically healthy
* At least 24 teeth in the functional dentition, excluding third molars
* Clinical diagnosis of periodontal health (no periodontal pockets > 3 mm, bleeding on probing percentage < 10%, and no attachment loss).

Exclusion criteria:

* Smokers.
* Medically compromised patients.
* Pregnant woman.
* Allergies to green tea or EO.
* Any condition that might affect the periodontal tissues.
* Patients with any carious lesions (initial or active).
* Patients who have overhang restorations, poorly designed crowns or bridges, and ortho retainers.
* Use of systemic antibiotics or anti-inflammatory medications within 3 months prior to enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Turesky modification of the Quigley-Hein plaque index (TM-QHPI) | On days 0, 7, 14, and 21
  will be recorded at six aspects on each tooth (mesialbuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual).
  0: No plaque.
  1. Separate flecks of plaque at the gumline (cervical margin).
  2. A thin, continuous band (up to 1 mm) at the gumline.
  3. A band wider than 1 mm but covering less than one-third of the tooth crown.
  4. Plaque covering one-third to two-thirds of the crown.
  5. Plaque covering two-thirds or more of the crown.

SECONDARY OUTCOMES:
Gingival Index (GI) | On days 0, 7, 14, and 21
  Gingival inflammation will be evaluated using the Löe & Silness Gingival Index (GI). It will be recorded at six aspects on each tooth (mesialbuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual).
  Gingival index 0: Healthy gums. Gingival index 1: Mild discolouration and oedematous gingiva. No bleeding on probing.
  Gingival index 2: Red, oedematous and shiny gingiva. There is bleeding on probing.
  Gingival index 3: Red, oedematous and ulcerated gingiva. There is spontaneous bleeding.
The Discoloration Index (DI) | On days 0, 7, 14, and 21
  will be recorded at six aspects on each tooth (mesialbuccal, midbuccal, distobuccal, mesiolingual, midlingual, and distolingual).
  Score 0: No discoloration, clean and polished tooth surface, natural appearance in color.
  Score1: Slight yellowing discoloration, yellowish film over the entire extent of the clinical crown, slight brownish discoloration along the gingival margin.
  Score 2: Moderate brownish discoloration on the interproximal surfaces and in the apical third of the clinical crown.
  Score 3: Heavy brown and black discoloration over the entire extent of the tooth surface, black discoloration predominantly on the interproximal surfaces
Patient-reported outcome | On days 7, 14, and 21
  A self-reported outcome assessing participants' perceived feeling of oral freshness, good breath and cleanliness after using the assigned mouthwash. Each participant will rate their experience on a Visual Analogue Scale (VAS) from 0 ("not fresh or clean at all") to 10 ("very fresh and clean").

CONTACTS AND LOCATIONS:
Overall Officials: Lana Bader, DClinDent Perio, Study Director — Jordan University of Science and Technology; Dana Abdullah, MClinDent Perio, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Faculty of Dentistry, Irbid, Irbid Governorate, Jordan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data for plaque index, gingival index, discolouration index, and patient-reported outcomes will be shared. Data will be stripped of all identifiers to protect participant privacy.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Individual Participant Data (IPD) and supporting documents (Study Protocol, Statistical Analysis Plan, Informed Consent Form, and Clinical Study Report) will be made available after publication of the study results, approximately one year after study completion.
Access Criteria: Access will be granted to qualified researchers who request the data via email to the principal investigator. Researchers must sign a data use agreement ensuring ethical use, confidentiality, and prohibition of attempts to identify participants.